CLINICAL TRIAL: NCT06231680
Title: A Prospective, Randomized Clinical Study of the Prevention or Treatment of Camrelizumab-induced Reactive Cutaneous Capillary Endothelial Proliferation (RCCEP) With Thalidomide
Brief Title: Thalidomide Prevention or Treatment of Camrelizumab-induced Reactive Cutaneous Capillary Endothelial Proliferation (RCCEP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Ying Liu, Deputy Chief Physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-RCCEP-II-001
Record Dates: First submitted 2023-11-07; First posted 2024-01-30 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer, Nonsmall Cell; Esophageal Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms | interventions — camrelizumab; Thalidomide; Drug Therapy; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prevention Cohort 1 Group A (Experimental): Camrelizumab + chemotherapy+Thalidomide(50mg)
  Interventions: Drug: Camrelizumab; Drug: Thalidomide 50mg; Drug: Chemotherapy
- Prevention Cohort 1 Group B (Experimental): Camrelizumab + chemotherapy+Thalidomide(100mg)
  Interventions: Drug: Camrelizumab; Drug: Thalidomide 100mg; Drug: Chemotherapy
- Treatment Cohort 2 Group A (Experimental): Thalidomide(100mg)
  Interventions: Drug: Thalidomide 100mg
- Treatment Cohort 2 Group B (Experimental): Thalidomide(200mg)
  Interventions: Drug: Thalidomide 200mg

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg intravenous (IV) on Day 1 of each 21-day cycle，until progression or unacceptable toxicity
  Other Names: SHR-1210
  Arms: Prevention Cohort 1 Group A; Prevention Cohort 1 Group B
Drug: Thalidomide 50mg — Thalidomide 50mg，po qd；
  Other Names: Thalidomide
  Arms: Prevention Cohort 1 Group A
Drug: Thalidomide 100mg — Thalidomide 100mg，po qd；
  Other Names: Thalidomide
  Arms: Prevention Cohort 1 Group B; Treatment Cohort 2 Group A
Drug: Thalidomide 200mg — Thalidomide 200mg，po qd；
  Other Names: Thalidomide
  Arms: Treatment Cohort 2 Group B
Drug: Chemotherapy — Platinum-based chemotherapy:
  1. Esophageal squamous cell carcinoma: cisplatin/carboplatin/nedaplatin/lobaplatin+ paclitaxel/albumin-bound paclitaxel/fluorouracil on Day 1 of each 21-day cycle for 4-6 cycles;
  2. Non-small cell lung cancer (non-squamous cell carcinoma): pemetrexed plus carboplatin/cisplatin on Day 1 of each 21-day cycle for 4-6 cycles，pemetrexed every three weeks (Q3W) maintenance for the remainder of the study or until documented PD;
  3. Non-small cell lung cancer (squamous cell carcinoma) : paclitaxel/albumin-bound paclitaxel + carboplatin/cisplatin on Day 1 of each 21-day cycle for 4-6 cycles.
  Other Names: Platinum-based chemotherapy
  Arms: Prevention Cohort 1 Group A; Prevention Cohort 1 Group B

SUMMARY:
To explore the dose and safety of thalidomide for the prevention and treatment of camrelizumab-induced reactive cutaneous capillary endothelial proliferation (RCCEP)

DETAILED DESCRIPTION:
1. To increase the evidence of thalidomide for the prevention of RCCEP, the investigators will explore the dose of thalidomide for the prevention of RCCEP in participants with esophageal squamous cell carcinoma and non-small cell lung cancer who were scheduled to receive camrelizumab combined with platinum-based chemotherapy;
2. To increase the evidence of thalidomide for the treatment of RCCEP, the investigators will explore the dose of thalidomide for the treatment of ≥G2 RCCEP in participants with esophageal squamous cell carcinoma and non-small cell lung cancer with camrelizumab

ELIGIBILITY:
Inclusion Criteria:

* Prevention cohort 1:

  1. Histopathology or cytology confirmed advanced non-small cell lung cancer or esophageal squamous cell carcinoma; no previous systemic therapy (patients who had progressed ≥6 months after [neo] adjuvant therapy were eligible).
  2. A treatment regimen of Camrelizumab combined with platinum-containing chemotherapy is planned.
  3. ECOG: 0-1;
  4. Age ≥18 years old;
  5. Have a life expectancy of at least 12 weeks;
  6. No prior therapy with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
  7. Can swallow pills normally;
  8. Adequate organ and bone marrow function：Standard of blood routine examination (without transfusion within 14 days) : Hemoglobin (HB) ≥80 g/L; Neutrophil absolute value (ANC) ≥1.5×10^9/L; Platelet (PLT) ≥90×10^9/L;Biochemical examination should meet the following criteria: Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤3×ULN; Serum creatinine (Cr) ≤1.5 ULN;
  9. Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 2 months after the last dose of study treatment. Male Subjects with a female partner(s) of child-bearing potential must be willing to use very efficient barrier methods of contraception for the course of the study through 2 months after the last dose of study treatment;
  10. Subjects has voluntarily agreed to participate by giving written informed consent/assent for the trial.
* Treatment cohort 2:

  1. Histopathology or cytology confirmed advanced lung cancer or esophageal carcinoma;
  2. Subjects had≥G2 grade RCCEP for the first time after treatment with a Camrelizumab based regimen;
  3. ECOG: 0-2;
  4. Age ≥18 years old;
  5. Have a life expectancy of at least 12 weeks;
  6. Can swallow pills normally;
  7. No ongoing grade 3 or higher adverse events except for RCCEP (according to CTCAE version 5.0).
  8. Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 2 months after the last dose of study treatment. Male Subjects with a female partner(s) of child-bearing potential must be willing to use very efficient barrier methods of contraception for the course of the study through 2 months after the last dose of study treatment;
  9. Subjects have voluntarily agreed to participate by giving written informed consent/assent for the trial.

Exclusion Criteria:

* Prevention cohort 1:

  1. Known allergy to the investigational drug or excipient, history of severe hypersensitivity reactions to other monoclonal antibodies.
  2. Subjects with a condition requiring systemic treatment with other immunosuppressive medications within 14 days of first administration of study treatment.
  3. Subjects had administration of a live, attenuated vaccine within 4 weeks of the first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study.
  4. Advanced patients who have symptoms, have spread to the internal organs, and are at risk of developing life-threatening complications in the short term;
  5. Subjects with a history of interstitial lung disease, or other disease may interfere with the detection or treatment of suspected drug-related lung toxicity.
  6. Subjects with active, known or suspected autoimmune disease. Subjects in conditions not expected to recur in the absence of an external trigger, or not requiring systemic treatment are permitted to enroll.
  7. HIV infection; Combined hepatitis B and hepatitis C co-infection
  8. Subjects with active CNS metastases are excluded.
  9. Subjects with clinically significant cardiovascular and cerebrovascular diseases.
  10. Coagulation abnormalities, with bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
  11. Disposition evidence of hemoptysis in 2 months (bright red blood, 1/2 teaspoon).
  12. History of hemorrhage within 3 months prior to the start of study treatment or clear tendency of hemorrhage
  13. Thrombosis or thromboembolic event within 6 months prior to the start of study treatment;
  14. Active infection (CTCAE> Grade 2)
  15. Subjects had or plan to have allogeneic bone marrow transplantation or solid organ transplant.
  16. Subjects are currently participating and receiving study therapy or had participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks or 5 half-value period life of the agent, before the first dose of trial treatment.
  17. Subjects have known psychiatric or substance abuse disorder
  18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Treatment cohort 2:

  1. Known allergy to the investigational drug or excipient
  2. Advanced patients who have symptoms, have spread to the internal organs, and are at risk of developing life-threatening complications in the short term;
  3. Subjects with a history of interstitial lung disease, or other disease may interfere with the detection or treatment of suspected drug-related lung toxicity.
  4. HIV infection; Combined hepatitis B and hepatitis C co-infection
  5. Active infection (CTCAE> Grade 2)
  6. Subjects have known psychiatric or substance abuse disorder
  7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of RCCEP | 2 years
  Incidence rate of RCCEP
RCCEP response rate at 3 weeks | 3 weeks
  RCCEP response rate at 3 weeks

SECONDARY OUTCOMES:
Incidence rate of ≥G3 grade RCCEP | 2 years
  Incidence rate of ≥G3 grade RCCEP
Median time to RCCEP | 2 years
  Median time to RCCEP
Incidence rate of RCCEP at 6 weeks | 6 weeks
  Incidence rate of RCCEP at 6 weeks
Incidence rate of RCCEP at 9 weeks | 9 weeks
  Incidence rate of RCCEP at 9 weeks
Median time to response of RCCEP | 2 years
  Median time to response of RCCEP
Thalidomide treatment-related adverse events | 2 years
  Thalidomide treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, MD, Principal Investigator — Henan Cancer Hospital; Yu Yao, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - Ying Liu, Zhengzhou, Henan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No